CLINICAL TRIAL: NCT01033942
Title: Acceptability and Feasibility of a Pre-Exposure Prophylaxis (PrEP) Trial With Young Men Who Have Sex With Men (YMSM)
Brief Title: Pre-Exposure Prophylaxis in YMSM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ATN 082
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Results first posted 2017-03-29 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-02

CONDITIONS: HIV
Keywords: Pre-exposure prophylaxis; HIV Prevention; Truvada; Many Men, Many Voices; Emtricitabine; Tenofovir disoproxil fumarate; Young men who have sex with men; HIV Seronegativity
MeSH Terms: interventions — Racivir; Tenofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- FTC/TDF as PrEP (Experimental): Blinded treatment with FTC (Emtricitabine) and TDf (Tenofovir)Pre-Exposure Prophylaxis (PrEP); HIV behavioral intervention
  Interventions: Drug: coformulated emtricitabine (FTC) and tenofovir disoproxil fumarate (TDF) as PrEP; Behavioral: Many Men, Many Voices (3MV)
- Placebo Pill Control (Placebo Comparator): Blinded administration of placebo pill; HIV behavioral intervention
  Interventions: Drug: Placebo; Behavioral: Many Men, Many Voices (3MV)
- No Pill Control (Active Comparator): Subjects receive HIV behavioral intervention but no pill.
  Interventions: Behavioral: Many Men, Many Voices (3MV)

INTERVENTIONS:
Drug: coformulated emtricitabine (FTC) and tenofovir disoproxil fumarate (TDF) as PrEP — Subjects receive PrEP and receive clinical follow-up visits every four weeks for 24 weeks.
  Arms: FTC/TDF as PrEP
Drug: Placebo — Subjects receive placebo and receive clinical follow-up visits every four weeks for 24 weeks.
  Arms: Placebo Pill Control
Behavioral: Many Men, Many Voices (3MV) — Behavioral HIV-prevention intervention. Behavioral and biomedical data will be collected at baseline and every 4 weeks thereafter for 24 weeks.

SUMMARY:
This is an exploratory mixed-methods research study that compares an efficacious behavioral HIV-prevention intervention (3MV) alone to the behavioral HIV-prevention intervention combined with a biomedical intervention (PrEP). After completing the 3MV behavioral intervention, participants will be randomly assigned to one of three study arms: 1) daily FTC/TDF as PrEP, 2) placebo pill control, or 3) "no pill" control. Behavioral and biomedical data will be collected at baseline and every 4 weeks thereafter for 24 weeks. Youth who decline to participate will be asked to complete a brief survey about their opinions on PrEP. Qualitative interviews will be completed with six study participants and the study coordinators at the end of the trial to explore further the issues of trial acceptability and feasibility. Finally, focus groups will be conducted to explore feasibility and acceptability issues with YMSM who meet all eligibility requirements of the study except for not being age 18 or older, but are at least 16 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to independently provide written informed consent;
* Of male gender at birth;
* Between the ages of 18 years and 0 days through 22 years and 364 days at the time of signed informed consent;
* Self-reporting at least one episode of unprotected anal intercourse with a male within the last 12 months at the time of Personal Digital Assistant (PDA) Screening Interview;
* Tests HIV negative at time of screening (using any FDA-approved HIV diagnostic test);
* Willing to provide locator information to study staff;
* Willing to be assigned to any of the three biomedical intervention conditions;
* Does not report intention to relocate out of the study area during the course of the study; and
* Does not have job/other obligations that would require long absences from the area (> 4 weeks at a time).

Exclusion Criteria:

* Transgender (behavioral intervention not targeted toward this population);
* Presence of serious psychiatric symptoms (e.g., active hallucinations);
* Visibly distraught at the time of consent (e.g., suicidal, homicidal, exhibiting violent behavior);
* Intoxicated or under the influence of alcohol or other drugs at the time of consent;
* Acute or chronic hepatitis B infection (exclude if hepatitis B surface antigen positive);
* Renal dysfunction (Creatinine Clearance < 75 ml/min); Use Cockcroft-Gault equation: Glomerular Filtration Rate (GFR) = (140-Age in years) x (Weight in kg) / (72 x serum creatinine) for males
* Any history of bone fractures not explained by trauma;
* Confirmed proteinuria (repeated positive [> 2+] urine dipstick), unless explained by orthostatic proteinuria;
* Confirmed glucosuria (repeated positive [> 1+] urine dipstick) in the presence of normal blood glucose (<120 mg/dL);
* Any Grade 3 toxicity on screening tests/assessments;
* Concurrent participation in an HIV vaccine study or other investigational drug study; or
* Known allergy/sensitivity to the study drug or its components.
* Use of disallowed medications

Ages: 18 Years to 22 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2009-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Principal Investigator — Adolescent Trials Network
Locations (2):
- United States (2):
  - Ruth M Rothstein CORE Center/ John H Stroger Jr Hospital, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois

REFERENCES:
- See also: Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN) Website — http://www.atnonline.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This research was conducted at two clinical sites in Chicago. Accrual was open between August 2009 and May 2011.
Pre-assignment Details: Young males were approached for screening in the community. If eligible, a clinic-based screening was done to confirm eligibility. If confirmed, participants attended a behavioral intervention. Then a week 0 was scheduled for randomization. 68 participants were enrolled; 10 discontinued prior to randomization, for a total of 58 participants.
Groups:
- FTC/TDF as PrEP: Blinded treatment with FTC (Emtricitabine) and Tenofovir (TDf) Pre-Exposure Prophylaxis (PrEP); HIV behavioral intervention
  Coformulated emtricitabine (FTC) and tenofovir disoproxil fumarate (TDF) as PrEP: Subjects receive PrEP and receive clinical follow-up visits every four weeks for 24 weeks.
  Many Men, Many Voices (3MV): Behavioral HIV-prevention intervention. Behavioral and biomedical data will be collected at baseline and every 4 weeks thereafter for 24 weeks.
Period: Overall Study
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Started | 20 | 19 | 19
Completed | 18 | 15 | 18
Not Completed | 2 | 4 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Enrolled in Extension Study | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control | Total
Number analyzed (Participants) | 20 | 19 | 19 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (1.44) | 20.26 (1.45) | 19.84 (0.96) | 19.97 (1.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 20 | 19 | 19 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 10 | 23
  Not Hispanic or Latino | 13 | 13 | 9 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 12 | 9 | 31
  White | 1 | 1 | 2 | 4
  More than one race | 8 | 6 | 8 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 19 | 19 | 58
Education [Number; unit: participants] — Not all participants answered every question.
  participants
    Eighth Grade of Less | 0 | 0 | 1 | 1
    GED | 0 | 1 | 1 | 2
    Highschool Diploma | 10 | 3 | 5 | 18
    Some College | 8 | 14 | 8 | 30
Current Employment [Number; unit: participants]
  Unemployed | 12 | 11 | 9 | 32
  Full Time | 2 | 2 | 2 | 6
  Part Time | 6 | 6 | 8 | 20
Housing Experience (Responded YES) [Number; unit: participants] — Not all participants answered every question
  participants
    Kicked out of House Due to Sexual Orientation | 4 | 2 | 3 | 9
    Spent at least 1 Night in Shelter S | 5 | 6 | 8 | 19
    Have Exchanged Sex for Money or Place to Stay | 2 | 3 | 5 | 10
Unprotected Anal Sex with Man in Past 30 Days [Number; unit: participants]
  Yes | 9 | 7 | 8 | 24
  No | 11 | 12 | 11 | 34
Unprotected Anal or Vaginal Sex with Woman [Number; unit: participants]
  Yes | 0 | 2 | 1 | 3
  No | 20 | 17 | 18 | 55

OUTCOME MEASURES:

1. Primary Outcome: Actual Number of Study Visits Completed by 24 Weeks
Description: This outcome measure looked at whether the actual number of study visits conducted by 24 weeks differed by treatment group over time.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: Visits
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
Visits | 3.5927 (0.7387) | 4.6263 (0.9783) | 4.6374 (0.9784)
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.6983, Chi-squared — The p-value is for the difference in treatment (TX) groups overall. The interaction between TX group and study time that tests whether the TX groups differed over time could not be tested due to small no. of subjects that missed visits during study

2. Secondary Outcome: Number of Participants Reporting No High-Risk Man With Man Sex Acts at Baseline
Description: A high-risk sex act was defined as an answer of greater than 0 to any of the following questions:
  With your male HIV positive male partners during the past month:
  How many times did you have insertive anal sex WITHOUT a condom? How many times did you have receptive anal sex WITHOUT a condom? How many times did you have insertive anal sex WITHOUT a condom? How many times did you have receptive anal sex WITHOUT a condom?
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants | 11 | 11 | 12
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.8722, Fisher Exact

3. Primary Outcome: Acceptability of Size of Pill
Time Frame: Week 24
Population: Not all participants answered every question and therefore the number of responses in the outcome measure data table does not match the number of participants analyzed.
Measure: Number; unit: Participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Participants
  Did not like it at all | 3 | 3
  Did not like | 3 | 3
  Liked | 3 | 6
  Liked a lot | 1 | 0
  Missing response | 10 | 7
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.6921, Fisher Exact — Not all subjects answered every question

4. Primary Outcome: Acceptability of the Taste of the Pill
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Did not like it at all | 4 | 3
  Did not like | 1 | 4
  Liked | 4 | 5
  Liked a lot | 1 | 0
  Missing response | 10 | 7
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.4655, Fisher Exact — Not all participants answered every question

5. Primary Outcome: Acceptability of the Color of the Pill
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Did not like it at all | 1 | 1
  Did not like | 2 | 3
  Liked | 4 | 5
  Liked a lot | 3 | 3
  Missing response | 10 | 7
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact — Not all participants answered every question

6. Primary Outcome: Acceptability of Taking the Pill Everyday
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Did not like it at all | 3 | 1
  Did not like | 3 | 7
  Liked | 2 | 4
  Liked a lot | 2 | 0
  Missing response | 10 | 7
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.2297, Fisher Exact — Not all participants answered every question

7. Primary Outcome: Acceptability of Taking Part in the Study
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like it at all | 2 | 0 | 0
  Did not like | 0 | 1 | 0
  Liked | 0 | 2 | 1
  Liked a lot | 8 | 9 | 12
  Missing response | 10 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1886, Fisher Exact — Not all participants answered every question

8. Primary Outcome: Acceptability of Participating in Group Sessions
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like it at all | 0 | 1 | 0
  Did not like | 1 | 2 | 0
  Liked | 0 | 2 | 4
  Liked a lot | 9 | 7 | 9
  Missing response | 10 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1908, Fisher Exact

9. Primary Outcome: Acceptability of Being Randomly Assigned to a Group
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like it at all | 1 | 4 | 0
  Did not like | 3 | 2 | 2
  Liked | 4 | 4 | 5
  Liked a lot | 1 | 2 | 6
  Missing response | 11 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2240, Fisher Exact — Not all participants answered every question

10. Primary Outcome: Acceptability of Having an HIV Test at Every Visit
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like | 0 | 1 | 0
  Liked | 0 | 3 | 1
  Liked a lot | 10 | 8 | 12
  Missing response | 10 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1538, Fisher Exact — Not all participants answered every question

11. Primary Outcome: Acceptability of Risk Reduction Counseling at Every Visit
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like it at all | 0 | 1 | 0
  Liked | 1 | 5 | 4
  Liked a lot | 9 | 6 | 9
  Missing response | 10 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2151, Fisher Exact — Not all participants answered every question

12. Primary Outcome: Acceptability of Questions About Sexual Behavior at Every Visit
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like it at all | 0 | 1 | 0
  Did not like | 0 | 1 | 0
  Liked | 1 | 4 | 4
  Liked a lot | 9 | 6 | 9
  Missing response | 10 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2809, Fisher Exact — Not all participants answered every question

13. Primary Outcome: Acceptability of Being Contacted by the Research Team in Between Visits
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like | 0 | 2 | 0
  Liked | 4 | 5 | 3
  Liked a lot | 6 | 4 | 10
  Missing response | 10 | 8 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1850, Fisher Exact — Not all participants answered every question

14. Primary Outcome: Acceptability of Physical Examination by a Doctor
Time Frame: Week 24
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like it at all | 0 | 3 | 0
  Did not like | 1 | 0 | 0
  Liked | 2 | 3 | 3
  Liked a lot | 7 | 6 | 10
  Missing response | 10 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2366, Fisher Exact — Not all participants answered every question

15. Primary Outcome: Acceptability of Health Clinic for Study Visits
Time Frame: Week 24
Population: Not all participants answered every question.
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants
  Did not like | 0 | 2 | 0
  Liked | 4 | 4 | 3
  Liked a lot | 6 | 6 | 10
  Missing response | 10 | 7 | 6
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.4089, Fisher Exact — Not all subjects answered every question

16. Primary Outcome: Number of Missed Doses Based on Self-Report Calendar Data-Week 4
Description: Missed doses were calculated as the number of days between the date that subject came in for their current visit and the last date the subject was dispensed medication minus the total number of days the subject records having taken their medication in the last 31 days based on self-report calendar data. Since each subject is given a 30 day supply of medication at each visit, any days after 30 days are assumed to be missed medication days and are included in the total. Participants were taking only one dose per day and thus, the number of missed doses is the same as the number of missed medication days.
Time Frame: 4 weeks
Measure: Median (Full Range); unit: Missed Doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed Doses | 10 [0 to 32] | 10 [0 to 27]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

17. Primary Outcome: Number of Missed Doses Based on Self-Report Calendar Data-Week 8
Description: as for outcome 16
Time Frame: Week 8
Measure: Median (Full Range); unit: Missed Doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed Doses | 14 [0 to 28] | 8 [0 to 29]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

18. Primary Outcome: Number of Missed Doses Based on Self-Report Calendar Data-Week 12
Description: as for outcome 16
Time Frame: Week 12
Measure: Median (Full Range); unit: Missed Doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed Doses | 10 [0 to 29] | 6.5 [0 to 28]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

19. Primary Outcome: Number of Missed Doses Based on Self-Report Calendar Data-Week 16
Description: as for outcome 16
Time Frame: Week 16
Measure: Median (Full Range); unit: Missed Doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed Doses | 5 [0 to 27] | 19 [0 to 28]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.7007, Fisher Exact

20. Primary Outcome: Number of Missed Doses Based on Self-Report Calendar Data-Week 20
Description: as for outcome 16
Time Frame: Week 20
Measure: Median (Full Range); unit: Missed Doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed Doses | 5 [0 to 35] | 10 [0 to 27]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

21. Primary Outcome: Number of Missed Doses Based on Self-Report Calendar Data-Week 24
Description: as for outcome 16
Time Frame: Week 24
Measure: Median (Full Range); unit: Missed Doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed Doses | 17 [0 to 35] | 5.5 [0 to 11]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

22. Primary Outcome: Number of Missed Doses Over Time Based on Self-Report Calendar Data
Description: The outcome measure presents the least square means from the generalized linear model. The outcome here is a binary variable that determines whether the subject missed a dose or not. In a binomial model with logit link, the least squares means are predicted population margins of the logits.
Time Frame: 24 weeks
Measure: Least Squares Mean (Standard Error); unit: Doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Doses | 0.4752 (0.3965) | 0.4021 (0.3596)
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.8934, Chi-squared

23. Primary Outcome: Number of Missed Doses Based on Medication Refill Dates-Week 4
Description: Missed doses were calculated as the number of days between the actual and expected refill dates. Participants were taking only one dose per day and thus, the number of missed doses is the same as the number of missed medication days.
Time Frame: Week 4
Measure: Median (Full Range); unit: Missed doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed doses | 0 [0 to 7] | 0 [0 to 2]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

24. Primary Outcome: Number of Missed Doses Based on Medication Refill Dates-Week 8
Description: as for outcome 23
Time Frame: Week 8
Measure: Median (Full Range); unit: Missed doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed doses | 0 [0 to 1] | 0 [0 to 3]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

25. Primary Outcome: Number of Missed Doses Based on Medication Refill Dates-Week 12
Description: as for outcome 23
Time Frame: Week 12
Measure: Median (Full Range); unit: Missed doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed doses | 0 [0 to 7] | 0 [0 to 1]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.9999, Fisher Exact

26. Primary Outcome: Number of Missed Doses Based on Medication Refill Dates-Week 16
Description: as for outcome 23
Time Frame: Week 16
Measure: Median (Full Range); unit: Missed doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed doses | 0 [0 to 8] | 0 [0 to 5]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.4003, Fisher Exact

27. Primary Outcome: Number of Missed Doses Based on Medication Refill Dates-Week 20
Description: as for outcome 23
Time Frame: Week 20
Measure: Median (Full Range); unit: Missed doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed doses | 0 [0 to 3] | 0 [0 to 8]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.6462, Fisher Exact

28. Primary Outcome: Number of Missed Doses Based on Medication Refill Dates-Overall
Description: as for outcome 23
Time Frame: 20 Weeks
Measure: Median (Full Range); unit: Missed doses
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
Missed doses | 0 [0 to 8] | 0 [0 to 8]
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.8505, Chi-squared

29. Primary Outcome: Percentage of Participants With Tenofovir Plasma Concentrations (mg/mL) Detected at Baseline
Description: Subjects reporting tenofovir is calculated as those subjects that had a tenofovir plasma concentration greater than zero (BLQ). Subjects with BLQ+ (<10 ng/mL) were included in this count.
Time Frame: Baseline
Population: Only two subjects in the Placebo Pill Control arm were randomly selected for tenofovir plasma concentration testing at baseline. All subjects in the FTC/TDF as PrEP arm had tenofovir plasma concentration testing and no subjects in the No Pill arm had tenofovir plasma concentration testing at baseline.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 2 | 0
percentage of participants | 0 | 0 |

30. Primary Outcome: Percentage of Participants With Tenofovir Plasma Concentrations (mg/mL) Detected at Week 4
Description: as for outcome 29
Time Frame: Week 4
Population: Only two subjects in the Placebo Pill Control arm were randomly selected for tenofovir plasma concentration testing at Week 4. 19 subjects in the FTC/TDF as PrEP arm had tenofovir plasma concentration testing and no subjects in the No Pill arm had tenofovir plasma concentration testing at Week 4.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 19 | 2 | 0
percentage of participants | 63.2 | 0 |

31. Primary Outcome: Percentage of Participants With Tenofovir Plasma Concentrations (mg/mL) Detected at Week 8
Description: as for outcome 29
Time Frame: Week 8
Population: 18 subjects in the Placebo Pill Control arm were randomly selected for tenofovir plasma concentration testing at Week 8. 17 subjects in the FTC/TDF as PrEP arm had tenofovir plasma concentration testing and 17 subjects in the No Pill arm had tenofovir plasma concentration testing at Week 8.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 17 | 18 | 17
percentage of participants | 47.1 | 0 | 0

32. Primary Outcome: Percentage of Participants With Tenofovir Plasma Concentrations (mg/mL) Detected at Week 12
Description: as for outcome 29
Time Frame: Week 12
Population: One subject in the Placebo Pill Control arm was randomly selected for tenofovir plasma concentration testing at Week 12. 15 subjects in the FTC/TDF as PrEP arm had tenofovir plasma concentration testing and 1 subject in the No Pill arm had tenofovir plasma concentration testing at Week 12.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 15 | 1 | 1
percentage of participants | 60 | 0 | 0

33. Primary Outcome: Percentage of Participants With Tenofovir Plasma Concentrations (mg/mL) Detected at Week 16
Description: as for outcome 29
Time Frame: Week 16
Population: 13 subjects in the Placebo Pill Control arm were randomly selected for tenofovir plasma concentration testing at Week 16. 13 subjects in the FTC/TDF as PrEP arm had tenofovir plasma concentration testing and 14 subjects in the No Pill arm had tenofovir plasma concentration testing at Week 16.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 13 | 13 | 14
percentage of participants | 53.8 | 0 | 0

34. Primary Outcome: Percentage of Participants With Tenofovir Plasma Concentrations (mg/mL) Detected at Week 20
Description: as for outcome 29
Time Frame: Week 20
Population: One subject in the Placebo Pill Control arm was randomly selected for tenofovir plasma concentration testing at Week 20. 12 subjects in the FTC/TDF as PrEP arm had tenofovir plasma concentration testing and no subjects in the No Pill arm had tenofovir plasma concentration testing at Week 20.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 12 | 1 | 0
percentage of participants | 41.7 | 0 |

35. Primary Outcome: Percentage of Participants With Tenofovir Plasma Concentrations (mg/mL) Detected at Week 24
Description: as for outcome 29
Time Frame: Week 24
Population: No subjects in the Placebo Pill Control arm were randomly selected for tenofovir plasma concentration testing at Week 24. 10 subjects in the FTC/TDF as PrEP arm had tenofovir plasma concentration testing and no subjects in the No Pill arm had tenofovir plasma concentration testing at Week 24.
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 10 | 0 | 0
percentage of participants | 20 |  |

36. Primary Outcome: Frequency of Missing Study Pills Because Participant Was Away From Home
Time Frame: 24 Weeks
Population: Participants in the No Pill Control arm were not included in the analysis. Analysis measure type is the percentage of participants in each frequency category for missed dose reason.
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 31.76 | 48.39 |
  Rarely | 34.12 | 20.43 |
  Sometimes | 16.47 | 26.88 |
  Often | 17.65 | 4.30 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.7434, Chi-squared

37. Primary Outcome: Frequency of Missing Study Pills Because Participant Was Too Busy With Other Things
Time Frame: 24 Weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 47.06 | 58.06 |
  Rarely | 30.59 | 16.13 |
  Sometimes | 15.29 | 21.51 |
  Often | 7.06 | 4.30 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.6153, Chi-squared

38. Primary Outcome: Frequency of Missing Study Pills Because Participant Simply Forgot
Time Frame: 24 Weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 38.82 | 60.22 |
  Rarely | 40.00 | 16.13 |
  Sometimes | 9.41 | 15.05 |
  Often | 11.76 | 8.60 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.2000, Chi-squared

39. Primary Outcome: Frequency of Missing Study Pills Because Participant Had Too Many Study Pills to Take
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 92.94 | 95.70 |
  Rarely | 7.06 | 2.15 |
  Sometimes | 0.00 | 1.08 |
  Often | 0.00 | 1.08 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.5265, Chi-squared

40. Primary Outcome: Frequency of Missing Study Pills Because Participant Wanted to Avoid Side Effects
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 82.35 | 91.40 |
  Rarely | 9.41 | 3.23 |
  Sometimes | 0.00 | 2.15 |
  Often | 8.24 | 3.23 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.2559, Chi-squared

41. Primary Outcome: Frequency of Missing Study Pills Because Participant Did Not Want Others to Notice Participant Was Taking Medications
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 88.24 | 92.47 |
  Rarely | 5.88 | 4.30 |
  Sometimes | 2.35 | 0.00 |
  Often | 3.53 | 3.23 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.3846, Chi-squared

42. Primary Outcome: Frequency of Missing Study Pills Because Participant Had a Change in Daily Routine
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 62.35 | 70.97 |
  Rarely | 25.53 | 15.05 |
  Sometimes | 7.06 | 10.75 |
  Often | 7.06 | 3.23 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.5133, Chi-squared

43. Primary Outcome: Frequency of Missing Pills Because Participant Felt Like the Study Pill Was Toxic/Harmful
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 87.06 | 95.70 |
  Rarely | 5.88 | 2.15 |
  Sometimes | 3.53 | 0.00 |
  Often | 3.53 | 2.15 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.1661, Chi-squared

44. Primary Outcome: Frequency of Missing Study Pills Because Participant Fell Asleep/Slept Through Dose Time
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 68.24 | 86.02 |
  Rarely | 24.71 | 6.45 |
  Sometimes | 4.71 | 4.30 |
  Often | 2.35 | 3.23 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.0729, Chi-squared

45. Primary Outcome: Frequency of Missing Study Pills Because Participant Felt Sick or Ill
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 81.18 | 89.25 |
  Rarely | 11.76 | 5.38 |
  Sometimes | 4.71 | 3.23 |
  Often | 2.35 | 2.15 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.1912, Chi-squared

46. Primary Outcome: Frequency of Missing Study Pills Because Participant Felt Depressed/Overwhelmed
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 83.53 | 92.47 |
  Rarely | 12.94 | 2.15 |
  Sometimes | 0.00 | 3.23 |
  Often | 3.53 | 2.15 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.2829, Chi-squared

47. Primary Outcome: Frequency of Missing Study Pills Because Participant Ran Out of Study Pills
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 94.12 | 97.85 |
  Rarely | 4.71 | 1.08 |
  Sometimes | 0.00 | 1.08 |
  Often | 1.18 | 0.00 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.2685, Chi-squared

48. Primary Outcome: Frequency of Missing Study Pills Because Participant Didn't Think it Was Needed Because he/She Was Not Engaged in Risky Sex
Time Frame: 24 weeks
Population: as for outcome 36
Measure: Number; unit: % of participants in each category
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 0
% of participants in each category
  Never | 90.59 | 96.77 |
  Rarely | 4.71 | 0.00 |
  Sometimes | 1.18 | 2.15 |
  Often | 3.53 | 1.08 |
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.2342, Chi-squared

49. Primary Outcome: Number of Participants Who Thought They Were on Placebo vs. Pre-Exposure Prophylaxis (PrEP) at Week 4
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Placebo | 9 | 10
  PrEP | 4 | 1
  Don't Know | 5 | 6
  Don't Understand Question | 1 | 1
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.7314, Fisher Exact

50. Primary Outcome: Number of Participants Who Thought They Were on Placebo vs. Pre-Exposure Prophylaxis (PrEP) at Week 8
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Placebo | 8 | 9
  PrEP | 5 | 2
  Don't Know | 4 | 7
  Don't Understand Question | 0 | 0
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.3770, Fisher Exact

51. Primary Outcome: Number of Participants Who Thought They Were on Placebo vs. Pre-Exposure Prophylaxis (PrEP) at Week 12
Time Frame: Week 12
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Placebo | 6 | 6
  PrEP | 3 | 2
  Don't Know | 5 | 8
  Don't Understand Question | 0 | 0
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.7004, Fisher Exact

52. Primary Outcome: Number of Participants Who Thought They Were on Placebo vs. Pre-Exposure Prophylaxis (PrEP) at Week 16
Time Frame: Week 16
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Placebo | 6 | 5
  PrEP | 2 | 1
  Don't Know | 4 | 9
  Don't Understand Question | 0 | 0
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.4668, Fisher Exact

53. Primary Outcome: Number of Participants Who Thought They Were on Placebo vs. Pre-Exposure Prophylaxis (PrEP) at Week 20
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Placebo | 4 | 6
  PrEP | 3 | 2
  Don't Know | 4 | 6
  Don't Understand Question | 0 | 0
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.7573, Fisher Exact

54. Primary Outcome: Number of Participants Who Thought They Were on Placebo vs. Pre-Exposure Prophylaxis (PrEP) at Week 24
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control
Number analyzed (Participants) | 20 | 19
participants
  Placebo | 2 | 8
  PrEP | 3 | 0
  Don't Know | 4 | 4
  Don't Understand Question | 0 | 0
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control; Test type: Superiority or Other; p = 0.0356, Fisher Exact

55. Primary Outcome: Perceived Risk of Becoming HIV Positive at Week 4
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "Because I am in this PrEP study, I am less concerned about becoming HIV positive".
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 52.63 | 38.89 | 33.33
  Disagree | 21.05 | 33.33 | 22.22
  Neutral | 10.53 | 11.11 | 27.78
  Agree | 15.79 | 11.11 | 0.00
  Strongly Agree | 0.00 | 5.56 | 16.67
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.3176, Fisher Exact

56. Primary Outcome: Perceived Risk of Becoming HIV Positive at Week 8
Description: as for outcome 55
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 29.41 | 66.67 | 58.82
  Disagree | 17.65 | 27.78 | 11.76
  Neutral | 23.53 | 0.00 | 11.76
  Agree | 23.53 | 5.56 | 11.76
  Strongly Agree | 5.88 | 0.00 | 5.88
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1348, Fisher Exact

57. Primary Outcome: Perceived Risk of Becoming HIV Positive at Week 12
Description: as for outcome 55
Time Frame: Week 12
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 40.00 | 75.00 | 31.25
  Disagree | 40.00 | 6.25 | 37.50
  Neutral | 20.00 | 6.25 | 12.50
  Agree | 0.00 | 12.50 | 6.25
  Strongly Agree | 0.00 | 0.00 | 12.50
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0420, Fisher Exact

58. Primary Outcome: Perceived Risk of Becoming HIV Positive at Week 16
Description: as for outcome 55
Time Frame: Week 16
Population: Not all participants answered every question
Measure: Number; unit: percentage of partcipants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of partcipants
  Strongly Disagree | 58.33 | 80.00 | 42.86
  Disagree | 16.67 | 13.33 | 21.43
  Neutral | 8.33 | 6.67 | 21.43
  Agree | 8.33 | 0.00 | 0.00
  Strongly Agree | 8.33 | 0.00 | 14.29
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.4906, Fisher Exact

59. Primary Outcome: Perceived Risk of Becoming HIV Positive at Week 20
Description: as for outcome 55
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 66.67 | 78.57 | 30.77
  Disagree | 16.67 | 21.43 | 23.08
  Neutral | 0.00 | 0.00 | 23.08
  Agree | 16.67 | 0.00 | 7.69
  Strongly Agree | 0.00 | 0.00 | 15.38
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0544, Fisher Exact

60. Primary Outcome: Perceived Risk of Becoming HIV Positive at Week 24
Description: as for outcome 55
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 60.00 | 75.00 | 38.46
  Disagree | 20.00 | 8.33 | 23.08
  Neutral | 0.00 | 16.67 | 15.38
  Agree | 10.00 | 0.00 | 7.69
  Strongly Agree | 10.00 | 0.00 | 15.38
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.5645, Fisher Exact

61. Primary Outcome: Perceived HIV Risk Reduction at Week 4: Willingness to Take a Chance of Getting HIV Infected Because Participating in This PrEP Study
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "I am more willing to take a chance of getting infected now that I am in this PrEP study".
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 84.21 | 83.33 | 94.44
  Disagree | 5.26 | 5.56 | 0.00
  Neutral | 10.53 | 0.00 | 5.56
  Agree | 0.00 | 5.56 | 0.00
  Strongly Agree | 0.00 | 5.56 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.7847, Fisher Exact

62. Primary Outcome: Perceived HIV Risk Reduction at Week 8: Willingness to Take a Chance of Getting HIV Infected Because Participating in This PrEP Study
Description: as for outcome 61
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 68.75 | 100.00 | 64.71
  Disagree | 25.00 | 0.00 | 29.41
  Neutral | 6.25 | 0.00 | 5.88
  Agree | 0.00 | 0.00 | 0.00
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0288, Fisher Exact

63. Primary Outcome: Perceived HIV Risk Reduction at Week 12: Willingness to Take a Chance of Getting HIV Infected Because Participating in This PrEP Study
Description: as for outcome 61
Time Frame: Week 12
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 60.00 | 93.75 | 68.75
  Disagree | 33.33 | 0.00 | 18.75
  Neutral | 6.67 | 6.25 | 12.50
  Agree | 0.00 | 0.00 | 0.00
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0945, Fisher Exact

64. Primary Outcome: Perceived HIV Risk Reduction at Week 16: Willingness to Take a Chance of Getting HIV Infected Because Participating in This PrEP Study
Description: as for outcome 61
Time Frame: Week 16
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 66.67 | 93.33 | 71.43
  Disagree | 25.00 | 6.67 | 7.14
  Neutral | 0.00 | 0.00 | 7.14
  Agree | 8.33 | 0.00 | 7.14
  Strongly Agree | 0.00 | 0.00 | 7.14
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.3884, Fisher Exact

65. Primary Outcome: Perceived HIV Risk Reduction at Week 20: Willingness to Take a Chance of Getting HIV Infected Because Participating in This PrEP Study
Description: as for outcome 61
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 91.67 | 92.86 | 61.54
  Disagree | 8.33 | 7.14 | 30.77
  Neutral | 0.00 | 0.00 | 7.69
  Agree | 0.00 | 0.00 | 0.00
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2235, Fisher Exact

66. Primary Outcome: Perceived HIV Risk Reduction at Week 24: Willingness to Take a Chance of Getting HIV Infected Because Participating in This PrEP Study
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "I am more willing to take a chance of getting infected now that I am in this PrEP study."
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 80.00 | 91.67 | 53.85
  Disagree | 20.00 | 0.00 | 23.08
  Neutral | 0.00 | 0.00 | 23.08
  Agree | 0.00 | 8.33 | 0.00
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0467, Fisher Exact

67. Primary Outcome: Perceived HIV Risk Reduction at Week 4: Less Worried About 'Slipping up' Now That PrEP May be Taken Prior to Unprotected Sex
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "I am a lot less worried about 'slipping up' now that PrEP may be taken prior to unprotected sex."
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 66.67 | 55.56 | 55.56
  Disagree | 5.56 | 27.78 | 11.11
  Neutral | 11.11 | 5.56 | 16.67
  Agree | 11.11 | 5.56 | 16.67
  Strongly Agree | 5.56 | 5.56 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.6331, Fisher Exact

68. Primary Outcome: Perceived HIV Risk Reduction at Week 8: Less Worried About 'Slipping up' Now That PrEP May be Taken Prior to Unprotected Sex
Description: as for outcome 67
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 47.06 | 66.67 | 35.29
  Disagree | 29.41 | 5.56 | 35.29
  Neutral | 17.65 | 27.78 | 11.76
  Agree | 5.88 | 0.00 | 17.65
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0948, Fisher Exact

69. Primary Outcome: Perceived HIV Risk Reduction at Week 12: Less Worried About 'Slipping up' Now That PrEP May be Taken Prior to Unprotected Sex
Description: as for outcome 67
Time Frame: Week 12
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 64.29 | 68.75 | 43.75
  Disagree | 0.00 | 12.50 | 18.75
  Neutral | 21.43 | 12.50 | 18.75
  Agree | 14.29 | 6.25 | 18.75
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.5826, Fisher Exact

70. Primary Outcome: Perceived HIV Risk Reduction at Week 16: Less Worried About 'Slipping up' Now That PrEP May be Taken Prior to Unprotected Sex
Description: as for outcome 67
Time Frame: Week 16
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 53.85 | 93.33 | 42.86
  Disagree | 15.38 | 0.00 | 42.86
  Neutral | 23.08 | 6.67 | 7.14
  Agree | 7.69 | 0.00 | 0.00
  Strongly Agree | 0.00 | 0.00 | 7.14
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0087, Fisher Exact

71. Primary Outcome: Perceived HIV Risk Reduction at Week 20: Less Worried About 'Slipping up' Now That PrEP May be Taken Prior to Unprotected Sex
Description: as for outcome 67
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 75.00 | 78.57 | 38.46
  Disagree | 25.00 | 7.14 | 15.38
  Neutral | 0.00 | 7.14 | 15.38
  Agree | 0.00 | 7.14 | 23.08
  Strongly Agree | 0.00 | 0.00 | 7.69
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1934, Fisher Exact

72. Primary Outcome: Perceived HIV Risk Reduction at Week 24: Less Worried About 'Slipping up' Now That PrEP May be Taken Prior to Unprotected Sex
Description: as for outcome 67
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 50.00 | 83.33 | 46.15
  Disagree | 30.00 | 16.67 | 15.38
  Neutral | 10.00 | 0.00 | 23.08
  Agree | 0.00 | 0.00 | 15.38
  Strongly Agree | 10.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2146, Fisher Exact

73. Primary Outcome: Perceived HIV Risk Reduction at Week 4: Less Worried About Having Unprotected Sex Due to the Availability of PrEP
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "The availability of PrEP makes me less worried about having unprotected sex."
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 63.16 | 66.67 | 55.56
  Disagree | 5.26 | 16.67 | 27.78
  Neutral | 10.53 | 5.56 | 5.56
  Agree | 21.05 | 11.11 | 5.56
  Strongly Agree | 0.00 | 0.00 | 5.56
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.5317, Fisher Exact

74. Primary Outcome: Perceived HIV Risk Reduction at Week 8: Less Worried About Having Unprotected Sex Due to the Availability of PrEP
Description: as for outcome 73
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 58.82 | 66.67 | 35.29
  Disagree | 17.65 | 11.11 | 23.53
  Neutral | 17.65 | 16.67 | 11.76
  Agree | 0.00 | 5.56 | 29.41
  Strongly Agree | 5.88 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1733, Fisher Exact

75. Primary Outcome: Perceived HIV Risk Reduction at Week 12: Less Worried About Having Unprotected Sex Due to the Availability of PrEP
Description: as for outcome 73
Time Frame: Week 12
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 73.33 | 81.25 | 43.75
  Disagree | 20.00 | 6.25 | 18.75
  Neutral | 6.67 | 6.25 | 25.00
  Agree | 0.00 | 0.00 | 12.50
  Strongly Agree | 0.00 | 6.25 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1747, Fisher Exact

76. Primary Outcome: Perceived HIV Risk Reduction at Week 16: Less Worried About Having Unprotected Sex Due to the Availability of PrEP
Description: as for outcome 73
Time Frame: Week 16
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 58.33 | 80.00 | 35.71
  Disagree | 33.33 | 6.67 | 21.43
  Neutral | 8.33 | 13.33 | 28.57
  Agree | 0.00 | 0.00 | 0.00
  Strongly Agree | 0.00 | 0.00 | 14.29
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1203, Fisher Exact

77. Primary Outcome: Perceived HIV Risk Reduction at Week 20: Less Worried About Having Unprotected Sex Due to the Availability of PrEP
Description: as for outcome 73
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 66.67 | 78.57 | 53.85
  Disagree | 25.00 | 14.29 | 23.08
  Neutral | 8.33 | 7.14 | 15.38
  Agree | 0.00 | 0.00 | 7.69
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.8243, Fisher Exact

78. Primary Outcome: Perceived HIV Risk Reduction at Week 24: Less Worried About Having Unprotected Sex Due to the Availability of PrEP
Description: as for outcome 73
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 50.00 | 83.33 | 53.85
  Disagree | 30.00 | 8.33 | 15.38
  Neutral | 10.00 | 8.33 | 15.38
  Agree | 10.00 | 0.00 | 15.38
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.6202, Fisher Exact

79. Primary Outcome: Perceived HIV Risk Reduction at Week 4: Less Concerned About Unprotected Anal Sex Because Participating in This PrEP Study
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "I am less concerned about having unprotected anal sex now that I am in this PrEP study."
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 57.89 | 66.67 | 50.00
  Disagree | 26.32 | 22.22 | 27.78
  Neutral | 15.79 | 5.56 | 16.67
  Agree | 0.00 | 5.56 | 0.00
  Strongly Agree | 0.00 | 0.00 | 5.56
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.8351, Fisher Exact

80. Primary Outcome: Perceived HIV Risk Reduction at Week 8: Less Concerned About Unprotected Anal Sex Because Participating in This PrEP Study
Description: as for outcome 79
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 47.06 | 83.33 | 35.29
  Disagree | 23.53 | 11.11 | 41.18
  Neutral | 23.53 | 5.56 | 23.53
  Agree | 0.00 | 0.00 | 0.00
  Strongly Agree | 5.88 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.0484, Fisher Exact

81. Primary Outcome: Perceived HIV Risk Reduction at Week 12: Less Concerned About Unprotected Anal Sex Because Participating in This PrEP Study
Description: as for outcome 79
Time Frame: Week 12
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 57.14 | 81.25 | 50.00
  Disagree | 28.57 | 12.50 | 18.75
  Neutral | 7.14 | 6.25 | 25.00
  Agree | 7.14 | 0.00 | 6.25
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.4207, Fisher Exact

82. Primary Outcome: Perceived HIV Risk Reduction at Week 16: Less Concerned About Unprotected Anal Sex Because Participating in This PrEP Study
Description: as for outcome 79
Time Frame: Week 16
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 75.00 | 80.00 | 42.86
  Disagree | 25.00 | 6.67 | 28.57
  Neutral | 0.00 | 13.33 | 14.29
  Agree | 0.00 | 0.00 | 7.14
  Strongly Agree | 0.00 | 0.00 | 7.14
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2187, Fisher Exact

83. Primary Outcome: Perceived HIV Risk Reduction at Week 20: Less Concerned About Unprotected Anal Sex Because Participating in This PrEP Study
Description: as for outcome 79
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 75.00 | 92.86 | 61.54
  Disagree | 16.67 | 7.14 | 23.08
  Neutral | 0.00 | 0.00 | 7.69
  Agree | 8.33 | 0.00 | 7.69
  Strongly Agree | 0.00 | 0.00 | 0.00
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.5369, Fisher Exact

84. Primary Outcome: Perceived HIV Risk Reduction at Week 24: Less Concerned About Unprotected Anal Sex Because Participating in This PrEP Study
Description: as for outcome 79
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 60.00 | 83.33 | 46.15
  Disagree | 40.00 | 16.67 | 15.38
  Neutral | 0.00 | 0.00 | 23.08
  Agree | 0.00 | 0.00 | 7.69
  Strongly Agree | 0.00 | 0.00 | 7.69
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.1524, Fisher Exact

85. Primary Outcome: Perceived HIV Risk Reduction at Week 4: Participant Has Already Risked Getting HIV Infected Through Unprotected Sex While on This PrEP Study
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "I have already risked getting infected with HIV through unsafe sex while I've been in this study."
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 63.16 | 50.00 | 44.44
  Disagree | 5.26 | 16.67 | 5.56
  Neutral | 10.53 | 0.00 | 22.22
  Agree | 21.05 | 27.78 | 22.22
  Strongly Agree | 0.00 | 5.56 | 5.56
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.4700, Fisher Exact

86. Primary Outcome: Perceived HIV Risk Reduction at Week 8: Participant Has Already Risked Getting HIV Infected Through Unprotected Sex While on This PrEP Study
Description: as for outcome 85
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 52.94 | 61.11 | 23.53
  Disagree | 5.88 | 11.11 | 17.65
  Neutral | 17.65 | 5.56 | 23.53
  Agree | 5.88 | 5.56 | 17.65
  Strongly Agree | 17.65 | 16.67 | 17.65
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.4686, Fisher Exact

87. Primary Outcome: Perceived HIV Risk Reduction at Week 12: Participant Has Already Risked Getting HIV Infected Through Unprotected Sex While on This PrEP Study
Description: Participants were asked to state whether or not they strongly disagreed, disagreed, were neutral, agreed, or strongly agreed with the following statement: "I have already risked getting infected with HIV through unsafe sex while I've been on this study."
Time Frame: Week 12
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 46.67 | 68.75 | 25.00
  Disagree | 13.33 | 6.25 | 25.00
  Neutral | 13.33 | 18.75 | 18.75
  Agree | 13.33 | 6.25 | 18.75
  Strongly Agree | 13.33 | 0.00 | 12.50
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.3791, Fisher Exact

88. Primary Outcome: Perceived HIV Risk Reduction at Week 16: Participant Has Already Risked Getting HIV Infected Through Unprotected Sex While on This PrEP Study
Description: as for outcome 85
Time Frame: Week 16
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 46.15 | 66.67 | 42.86
  Disagree | 15.38 | 6.67 | 14.29
  Neutral | 15.38 | 6.67 | 7.14
  Agree | 7.69 | 20.00 | 21.43
  Strongly Agree | 15.38 | 0.00 | 14.29
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.7374, Fisher Exact

89. Primary Outcome: Perceived HIV Risk Reduction at Week 20: Participant Has Already Risked Getting HIV Infected Through Unprotected Sex While on This PrEP Study
Description: as for outcome 85
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 75.00 | 71.43 | 61.54
  Disagree | 8.33 | 21.43 | 15.38
  Neutral | 8.33 | 0.00 | 7.69
  Agree | 0.00 | 7.14 | 7.69
  Strongly Agree | 8.33 | 0.00 | 7.69
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.9363, Fisher Exact

90. Primary Outcome: Perceived HIV Risk Reduction at Week 24: Participant Has Already Risked Getting HIV Infected Through Unprotected Sex While on This PrEP Study
Description: as for outcome 85
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: percentage of participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
percentage of participants
  Strongly Disagree | 50.00 | 66.67 | 30.77
  Disagree | 10.00 | 16.67 | 15.38
  Neutral | 10.00 | 8.33 | 15.38
  Agree | 10.00 | 8.33 | 30.77
  Strongly Agree | 20.00 | 0.00 | 7.69
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.6267, Fisher Exact

91. Secondary Outcome: Number of Participants Reporting No High-Risk Man With Man Sex Acts at Week 4
Description: as for outcome 2
Time Frame: Week 4
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants | 15 | 14 | 12
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.6434, Fisher Exact

92. Secondary Outcome: Number of Participants Reporting No High-Risk Man With Man Sex Acts at Week 8
Description: as for outcome 2
Time Frame: Week 8
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants | 10 | 12 | 10
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.8582, Fisher Exact

93. Secondary Outcome: Number of Participants Reporting No High-Risk Man With Man Sex Acts at Week 12
Description: as for outcome 2
Time Frame: Week 12
Population: Not all participants answered every question.
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants | 13 | 14 | 12
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.5778, Fisher Exact

94. Secondary Outcome: Number of Participants Reporting No High-Risk Man With Man Sex Acts at Week 16
Description: as for outcome 2
Time Frame: Week 16
Population: Not all participants answered every question.
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants | 11 | 13 | 12
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.9881, Fisher Exact

95. Secondary Outcome: Number of Participants Reporting No High-Risk Man With Man Sex Acts at Week 20
Description: as for outcome 2
Time Frame: Week 20
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants | 9 | 11 | 10
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.9771, Fisher Exact

96. Secondary Outcome: Number of Participants Reporting No High-Risk Man With Man Sex Acts at Week 24
Description: as for outcome 2
Time Frame: Week 24
Population: Not all participants answered every question
Measure: Number; unit: participants
Arm/Group | FTC/TDF as PrEP | Placebo Pill Control | No Pill Control
Number analyzed (Participants) | 20 | 19 | 19
participants | 9 | 7 | 10
Statistical Analysis 1: Comparison: FTC/TDF as PrEP vs Placebo Pill Control vs No Pill Control; Test type: Superiority or Other; p = 0.2301, Fisher Exact

ADVERSE EVENTS:
Time Frame: 24 weeks
Groups:
- FTC/TDC: Blinded treatment with FTC (Emtricitabine) and TDf (Tenofovir)Pre-Exposure Prophylaxis (PrEP); HIV behavioral intervention
  Coformulated emtricitabine (FTC) and tenofovir disoproxil fumarate (TDF) as PrEP: Subjects receive PrEP and receive clinical follow-up visits every four weeks for 24 weeks.
  Many Men, Many Voices (3MV): Behavioral HIV-prevention intervention. Behavioral and biomedical data will be collected at baseline and every 4 weeks thereafter for 24 weeks.
- Placebo: Blinded administration of placebo pill; HIV behavioral intervention
  Placebo: Subjects receive placebo and receive clinical follow-up visits every four weeks for 24 weeks.
  Many Men, Many Voices (3MV): Behavioral HIV-prevention intervention. Behavioral and biomedical data will be collected at baseline and every 4 weeks thereafter for 24 weeks.
Arm/Group | FTC/TDC | Placebo | No Pill Control
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 4/20 | 1/19 | 0/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FTC/TDC (N=20) | Placebo (N=19) | No Pill Control (N=19)
Blood Bilirubin Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Protein Urine Present (Investigations) | 1 (1) | 0 (0) | 0 (0) — Grade 2
Creatinine Renal Clearance Decreased (Investigations) | 1 (2) | 0 (0) | 0 (0) — Grade 3
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Grade 3
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 4

LIMITATIONS AND CAVEATS:
After release of Pre-exposure Prophylaxis Initiative efficacy results, the Data and Safety Monitoring Board recommended that subjects be unblinded, enrollment stopped, all be offered option of PrEP, subjects on PrEP arm continued as scheduled.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Adolescent Medicine Trials Network (ATN) for HIV/AIDS Interventions Publication Policy outlines procedures for the development and review of abstracts, publications and presentations. The Adolescent Medicine Leadership Group (AMLG) retains custody of and primary rights to the data. Use of data must be approved by the protocol team and AMLG.